CLINICAL TRIAL: NCT02342132
Title: A Comparison of Three Methods for Improving Expiratory Cough Flow and Lung Volume in Children With Neuromuscular Diseases
Brief Title: Methods to Improve Expiratory Cough Flow and Lung Volume in Children With NMDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Seear, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H14-00473
Record Dates: First submitted 2014-07-25; First posted 2015-01-19 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Respiratoy Therapy Devices (Experimental): Non-Invasive Bipap Ventilator, Mechanical Insufflator-Exsufflator, and High Frequency Percussive Oscillator are the three respiratory therapy devices that all participants will be using in a random order, in three consecutive days, one device per day.
  Interventions: Device: Non-invasive bipap ventilator; Device: Mechanical insufflator-exsufflator; Device: High frequency percussive oscillator

INTERVENTIONS:
Device: Non-invasive bipap ventilator — The non-invasive bipap ventilator will be used in the following respiratory treatment: bipap assisted inspiratory breaths (BAIB). The patient will be encouraged to take deep breaths at least 1.5 times greater than resting tidal volume. The pressure assistance provided by the bipap starts at 10cm H2O. Patients already on bipap will use their home settings. Starting pressure is then increased as necessary to meet the maximal inspiratory goal volume in steps of 2 up to a maximum 20cm H2O. Once the ideal pressure of support levels are established, the child will perform 3 cycles of 5 deep breaths. After each cycle the patient will pause and perform huffing and assisted coughing. The patient will be suctioned as necessary.
Device: Mechanical insufflator-exsufflator — A commercial mechanical insufflator-exsufflator will be used in the following treatment: Mechanical insufflation-exsufflation (MI-E). The pressure will be administered by a face mask. The optimal pressure for the test will start at 10 cm H2O and will in crease in steps of 5 to a maximum of 25 cm H2O. The insufflation phase will take 3 seconds followed by a 2 second exsufflation phase. Three cycles of treatment will be used. Between each cycle the subject will pause and perform huffing and assisted coughing. The patient will be suctioned as necessary.
Device: High frequency percussive oscillator — A commercial high frequency percussive oscillator will be used in the following treatment: combined oscillation and nebulisation. Pressures will be delivered by a face mask. At higher oscillation frequencies it is usually necessary to support the cheeks. Pressure will be gradually be increased to accustom the child to a maximum of 25cm H2O. This standard maximal pressure will ideally be used for every child. A treatment cycle will consist of 3 minutes at a frequency of 2 Hz and pressure of 15cm H2O followed by 3 minutes of 4 Hz at 20cm H2O, then 3 minutes of 5 Hz at 25cm H2O. Throughout each cycle, the patient will receive nebulized saline through the machine. After each cycle the patient will pause and perform huffing and assisted coughing. The patient will be suctioned as necessary.

SUMMARY:
Children with neuromuscular diseases (NMDs) and weak chest muscles suffer frequent chest infections, hospital admissions and reduced life expectancy. Physiotherapy is widely used but there is limited research data to support choice of therapy. The investigators will study the clinical value of the three most commonly used chest physiotherapy devices in children with NMD's by measuring lung function tests before and after each of the three treatments. This is a pilot study. The best device will be selected for a long term study of early physiotherapy intervention in children with NMDs.

The treatments that have been developed to break the cycle of decreasing lung volume and poor secretion clearance, in children with NMDs, are all based on the same logical but unproved theory of treatment:

1. The loss of lung volume is reversed by applying positive pressure to the lungs via a face mask - literally reinflating the lungs with pressure. The three devices the investigators will test all provide positive pressure assistance during the inspiratory phase.
2. The temporarily increased lung volume then allows higher expiratory flow rates which helps to clear secretions. The expiratory phase is assisted by manual chest compression or, in one device, helped by application of negative pressure during exhalation.

All three devices that the investigators wish to compare follow this two-step approach. The hypotheses behind our study are:

1. Treatments combining positive pressure inhalation with assisted coughing during exhalation, will produce measurable improvements in lung volume and expiratory cough flow rates when tested in children with NMDs.
2. One of the three devices tested will be superior to the others. This will provide research-based justification for a long term study of the value of early intervention in children with NMDs.

DETAILED DESCRIPTION:
Current options for respiratory care in children with NMDs include numerous devices and treatments have been proposed for improving secretion clearance and lung function in very weak patients. Unfortunately treatment decisions are still based on little more than personal opinion. In particular, there are almost no carefully conducted studies on the best forms of respiratory therapy in children with NMDs. Commonly used treatment options are best listed under the following headings:

1. Chest physiotherapy. This broad term covers a range of therapies that includes postural drainage, manual percussion and chest vibrations. These treatments are often preceded by inhaled medications intended to mobilize secretions (humidification, hypertonic saline, Dornase alpha). Chest physiotherapy has been studied extensively in cystic fibrosis(13) but there are no prospective studies of its use in children with NMDs. The lack of any evidence of clear long-term benefit combined with the need for a trained assistant, has limited the application of chest therapy to in-patient treatment of acute exacerbations.
2. Breath stacking. Inspiratory lung volume can be increased by 'stacking' repeated inhalations. This allows a greater cough flow with improved secretion clearance. The simplest method is to use a bag, face mask and a one-way valve. Inspiratory volume can also be augmented using mechanical or non-invasive ventilators although care must be taken to avoid over-inflation and barotrauma(14). The cough phase after insufflation is often augmented by external compression of chest or abdomen (manually assisted cough). While there is evidence that breath stacking, with or without manually assisted coughing, can increase lung volume and peak cough flows(15), there are no prospective studies to study long term effects.
3. Mechanical insufflation-exsufflation. Devices in this group inflate the lung with an inspiratory positive pressure phase followed rapidly by a negative pressure exhalation phase(16). They are widely used and recommended but prospective research support is lacking. As with breath stacking, there is evidence of short term improvement in lung volume and cough flows(17) following MI-E treatment. There are also retrospective reviews to suggest that the technique is effective and well tolerated in children(18). However, there are no prospective controlled studies of MI-E either in adults or children.
4. Airway oscillation. Various devices have been developed to superimpose an oscillatory wave flow over normal breathing. The oscillating pressure wave is intended to help mobilise secretions and expand atelectatic areas of the lung. This can be achieved by an external vibrating vest or delivered directly to the airway through a face mask. Prospective study of the vibrating vest showed that it had no benefit(19). However, research exists that oscillation via mask is beneficial both in short(20) and longer term studies(21).

The newcomer to this important topic would be forgiven for finding the lack of research evidence difficult to believe. Children with NMDs are very complex management problems and they consume a lot of hospital resources. The mechanical devices paid for by insurance companies, or governments, cost many thousands of dollars each - surely all this money and time should be based on some form of evidence? Unfortunately this is not the case. Two large reviews of the management of NMDs by both the British(2) and the American(22) thoracic societies emphasized this lack of evidence. Both concluded that the major requirement in the management of these children is research.

The principal question in the management of children with NMDs is whether early introduction of effective respiratory therapy will slow the decline in lung function and help to keep these children out of hospital. That requires long term studies of the use of therapies known to be effective, at least in the short term. Such evidence - even short term evidence of efficacy, is not available. Our study is not a case of comparing a new treatment to an established therapy, it is a case of assessing current widely used treatments in order to determine whether they have any measurable benefits. The best of the three techniques studied will then form the basis for a long term early intervention study.

OBJECTIVES.

The short, medium and long term objectives of the study are as follows:

1. Short term objective.

   The principal short term aims are to answer the following research questions:
   * Do positive pressure reparatory physiotherapy devices increase lung volume and peak cough flows in children with neuromuscular diseases?
   * If there is a measurable effect on lung mechanics, which of the three most commonly used devices produces the biggest benefit?
2. Medium term objective. Assuming the investigators can show that one of the three devices has a significant beneficial short term effect on lung mechanics, the investigators will use that device in a much longer term study. This will investigate the possibility that early intervention with effective physiotherapy will slow the decline in lung function in children with NMDs. This is one of the main questions in the management of children with NMDs and it has never been addressed.
3. Long term objective. This proposal is the third in our series of planned studies on children with NMDs. Our long term objective is to help base the management of patients with this group of diseases on a firm research basis.

RESEARCH METHOD. Patient recruitment. Patients enrolled in the NMD clinic at children's hospital will initially be informed about the study by letter signed by the director of the NMD clinic, Dr Selby. At their next routine clinic visit, they will be approached by one of the two PIs (Dr Seear or Dr Selby). They will be given more information about the study and a handout covering the details. Once they have had time to consider the information, they will be invited to enroll in the study.

Patient eligibility. The study is open to children with neuro-muscular diseases of any type, who are enrolled in the NMD clinic at children's hospital. The main end points will be lung function measurements so children will need to be old enough to perform the testing process. For cognitively normal children this is usually 5 to 6 yrs of age. All of the three treatments are administered by a face mask so, apart from lack of consent and clinical instability, the only other exclusion criteria will be factors that limit the use of a face mask. Those children with a poor mask seal due to facial structural abnormalities, or those with tracheostomies will be ineligible for the study

General study design. After enrolment from the NMD clinic, children will be studied in batches of 15. Each batch will be studied over three consecutive weekdays so they can all receive the three treatments. On each of the study days, the group of fifteen will be randomized in groups of five to receive one of the three physiotherapy treatments. Each participant will receive all treatments at the end of the study and subsequently are considered one group. Randomization removes the chance of seeing an effect that may be due to a combination and not an individual treatment. Before and after each of the treatments, lung function tests will be measured by study staff blinded to the type of treatment. The respiratory function tests made before and after each treatment will be the same for each of the devices. By the end of the study period for that batch, every child will have completed three treatments.

Study treatment protocols.

In the absence of detailed research studies, there are no widely accepted protocols governing the three study treatments. After discussion with physiotherapy and respiratory technicians, the investigators have designed the three study protocols so they are representative of accepted common practice. Each treatment will be administered by a qualified physiotherapist who is familiar with the clinical use of the machine. The treatment will also be monitored by a physician in each of the three treatment rooms. Each child will receive the following study treatments in random order over three consecutive weekdays:

Measured end points. The effects of the three respiratory treatments will be assessed using standard lung function tests. A baseline will be obtained prior to each treatment. Repeat tests will be performed immediately after the treatment, then at ½, 1 and 2 hours later. Comparative predictive lung function values are based on algorithms that rely on patient height. In those children with severe spinal deformity, arm span will be used as a surrogate for height. All tests will be made by qualified respiratory technicians using regularly maintained and calibrated equipment. The staff measuring, reporting and storing the results will be blinded to the child's therapy. Other tests commonly used in the assessment of children with NMDs, such as oximetry and capnography, will not be measured since it is unlikely they will change over the short duration of the study. The following end points will be measured: lung volume, cough expiratory flows, and muscle strength.

STATISTICAL ANALYSIS. Measured endpoints. There are 4 measured endpoints: vital capacity (FVC in mls), peak expiratory flows (PEF in L/min), plus maximal inspiratory and expiratory pressures (MIP and MEP in cm H2O). All are continuous variables so will be expressed as mean+/- one standard deviation. Apart from graphical presentation of the results, the only statistical test will be a comparison of pre-treatment and post treatment values for each of the four variables.

Sample size. Before undertaking a long term study of early intervention with one of these three devices, the investigators would like to be at least 80% sure that they have a device that is able to produce a significant improvement in lung mechanics (20% improvement in post treatment mechanics). There are over a hundred types of NMD in children and the investigators will be testing the treatment effects of three devices. Unfortunately, there is currently no reliable evidence for the magnitude (or even existence) of any treatment effect and also the standard deviation of any effect. There is also no evidence of treatment variation when used in different sub-types of NMD. There is no basic data upon which to base a calculation of sample size. The investigators would have to make so many guesses that the calculated number would have no reliability. Our only response can be to try to enroll as many children as possible. There are over 200 children in the NMD clinic. The investigators hope to be able to enroll at least 100 of them.

Statistical tests. Any treatment effect will be detected by comparing baseline lung function tests to the post treatment values measured at 0, 1/2, 1 and 2 hours after the end of treatment. Each child's baseline values will serve as their own controls. Multiple comparisons of pre and post values will be made using Analysis of Variance with a Tukey post-hoc test.

ELIGIBILITY:
Inclusion Criteria:

* Child must have neuromuscular disease (of any diagnostic type)
* Child and family must be enrolled in the NMD clinic at Children's hospital
* Child must be old enough and cognitively able to perform lung function tests(usually about 5 to 6 years old)

Exclusion Criteria:

* Child or guardian refuses consent for the study
* Child has a tracheostomy
* Child is too young or cognitively unable to perform lung function tests
* Child has a facial asymmetry that prevents a good seal with the mask

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Lung Volume | Therapy effect assessed for 2hrs post treatment
  Assessed by measuring vital capacity (FVC). This is a widely used test that measures effective lung volume. There are well established pediatric predictive values for FVC.
Cough Expiratory Flows | Therapy effect assessed for 2hrs post treatment
  Cough flows needed for adequate clearance of airway secretions. This study will measure peak expiatory flow (PEF) for which normal values are easily accessible. The two measures are comparable in clinical use (8).
Muscle Strength | Therapy effect assessed for 2hrs post treatment
  Assessed by measuring maximal inspiratory pressure (MIP) and maximal expiratory pressures (MEP). These are obtained by inhaling and exhaling maximally through a manometer.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Seear, MD, Principal Investigator — British Columbia's Children's Hospital; Mike Seear, MD, Principal Investigator — BCCH
Locations (1):
- BC's Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Hull J, Aniapravan R, Chan E, Chatwin M, Forton J, Gallagher J, Gibson N, Gordon J, Hughes I, McCulloch R, Russell RR, Simonds A. British Thoracic Society guideline for respiratory management of children with neuromuscular weakness. Thorax. 2012 Jul;67 Suppl 1:i1-40. doi: 10.1136/thoraxjnl-2012-201964. No abstract available. PMID 22730428
- [Background] Suarez AA, Pessolano FA, Monteiro SG, Ferreyra G, Capria ME, Mesa L, Dubrovsky A, De Vito EL. Peak flow and peak cough flow in the evaluation of expiratory muscle weakness and bulbar impairment in patients with neuromuscular disease. Am J Phys Med Rehabil. 2002 Jul;81(7):506-11. doi: 10.1097/00002060-200207000-00007. PMID 12131177
- [Background] McCool FD, Rosen MJ. Nonpharmacologic airway clearance therapies: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):250S-259S. doi: 10.1378/chest.129.1_suppl.250S. PMID 16428718
- [Background] Jenkins HM, Stocki A, Kriellaars D, Pasterkamp H. Breath stacking in children with neuromuscular disorders. Pediatr Pulmonol. 2014 Jun;49(6):544-53. doi: 10.1002/ppul.22865. Epub 2013 Aug 16. PMID 23956183
- [Background] Toussaint M, Boitano LJ, Gathot V, Steens M, Soudon P. Limits of effective cough-augmentation techniques in patients with neuromuscular disease. Respir Care. 2009 Mar;54(3):359-66. PMID 19245730
- [Background] Homnick DN. Mechanical insufflation-exsufflation for airway mucus clearance. Respir Care. 2007 Oct;52(10):1296-305; discussion 1306-7. PMID 17894900
- [Background] Chatwin M, Ross E, Hart N, Nickol AH, Polkey MI, Simonds AK. Cough augmentation with mechanical insufflation/exsufflation in patients with neuromuscular weakness. Eur Respir J. 2003 Mar;21(3):502-8. doi: 10.1183/09031936.03.00048102. PMID 12662009
- [Background] Miske LJ, Hickey EM, Kolb SM, Weiner DJ, Panitch HB. Use of the mechanical in-exsufflator in pediatric patients with neuromuscular disease and impaired cough. Chest. 2004 Apr;125(4):1406-12. doi: 10.1378/chest.125.4.1406. PMID 15078753
- [Background] McIlwaine MP, Alarie N, Davidson GF, Lands LC, Ratjen F, Milner R, Owen B, Agnew JL. Long-term multicentre randomised controlled study of high frequency chest wall oscillation versus positive expiratory pressure mask in cystic fibrosis. Thorax. 2013 Aug;68(8):746-51. doi: 10.1136/thoraxjnl-2012-202915. Epub 2013 Feb 13. PMID 23407019
- [Background] Toussaint M, De Win H, Steens M, Soudon P. Effect of intrapulmonary percussive ventilation on mucus clearance in duchenne muscular dystrophy patients: a preliminary report. Respir Care. 2003 Oct;48(10):940-7. PMID 14525630
- [Background] Reardon CC, Christiansen D, Barnett ED, Cabral HJ. Intrapulmonary percussive ventilation vs incentive spirometry for children with neuromuscular disease. Arch Pediatr Adolesc Med. 2005 Jun;159(6):526-31. doi: 10.1001/archpedi.159.6.526. PMID 15939850
- [Background] Finder JD, Birnkrant D, Carl J, Farber HJ, Gozal D, Iannaccone ST, Kovesi T, Kravitz RM, Panitch H, Schramm C, Schroth M, Sharma G, Sievers L, Silvestri JM, Sterni L; American Thoracic Society. Respiratory care of the patient with Duchenne muscular dystrophy: ATS consensus statement. Am J Respir Crit Care Med. 2004 Aug 15;170(4):456-65. doi: 10.1164/rccm.200307-885ST. No abstract available. PMID 15302625